CLINICAL TRIAL: NCT05798221
Title: Complementary Self-help Strategies for Patients With Post-COVID-19 Syndrome: A Randomized Controlled Trial
Brief Title: Complementary Self-help Strategies for Patients With Post-COVID-19 Syndrome
Acronym: NASH-POCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Heidemarie Haller, Principal Investigator, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-11002-BO
Record Dates: First submitted 2023-04-02; First posted 2023-04-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Post-COVID-19 Syndrome
Keywords: complementary medicine; COVID-19; post-COVID-19 Syndrome; randomized controlled trial; self-help
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complementary self-help strategies in addition to treatment as usual (Experimental): The experimental group consists of 10 weeks of group treatments with educative and actively practicing elements. The patients will also receive a booklet with self-help basics and descriptions of the techniques, which should facilitate the correct practice at home. Parallel treatment as usual is allowed.
  Interventions: Behavioral: Complementary self-help strategies in addition to treatment as usual
- Treatment as usual (Active Comparator): The active control group consists a 16-week waiting period, where treatment as usual is allowed. In case of acute worsening/progression of the symptoms, consultations with the study physician are offered anytime. After the waiting period, the control group will be offered the same units as in the experimental group.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Complementary self-help strategies in addition to treatment as usual — The 10-week group program consists of self-help strategies from complementary medicine approaches of TEM (Traditional European Medicine), TCM (Traditional Chinese Medicine), and TIM (Traditional Indian Medicine) in addition to treatment as usual
  Arms: Complementary self-help strategies in addition to treatment as usual
Other: Treatment as usual — The active control group consists a 16-week waiting period, where treatment as usual is allowed. In case of acute worsening/progression of the symptoms, consultations with the study physician are offered anytime. After the waiting period, the control group will be offered the same units as in the experimental group.
  Arms: Treatment as usual

SUMMARY:
Individuals affected by SARS-CoV-2 infection may subsequently be affected by the so-called post-COVID syndrome. The aim of the present study is to investigate the effects of a multimodal 10-week group program consisting of self-help strategies based on complementary medicine approaches of TEM (Traditional European Medicine), TCM (Traditional Chinese Medicine), and TIM (Traditional Indian Medicine) in addition to treatment as usual versus treatment as usual alone (no active study intervention/waiting list). Endpoints of the study include subjective quantitative and qualitative as well as objective (physician-reported) variables.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and older
* Confirmed COVID-19 diagnosis by: 1. polymerase chain reaction (PCR) test or 2. physician's letter/medical certificate/quarantine order due to ICD-10-GM U07.1 G or ICD-10-GM U09.9 G
* Sequelae symptoms, new symptoms/disabilities, or worsening of a pre-existing medical condition that occurred in the first 3 months after confirmed SARS-CoV-2 infection and persisted for more than 2 months
* At least 8 points (moderate symptom burden) out of a possible 32 points on the Somatic Symptom Scale-8 (SSS-8)

Exclusion Criteria:

* Patients who were treated with invasive ventilation during active SARS-CoV-2 infection
* Severe comorbid mental illness (e.g. addiction diagnosis, major depression) or other severe comorbid somatic illness (e.g. cancer without remission, severe pre-existing cardiovascular disease, insufficiency of other organs such as kidney or liver, acute febrile infection, other severe neurologic disease)
* Pregnancy or lactation
* Current pension application
* Simultaneous participation in other clinical/interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Post-COVID-19 symptom burden | Week 16
  Somatic Symptom Scale-8 (SSS-8): self-report scale from 0 to 32 points with higher scores indicating higher level of burden

SECONDARY OUTCOMES:
Post-COVID-19 symptom burden | Week 10
  Somatic Symptom Scale-8 (SSS-8): self-report scale from 0 to 32 points with higher scores indicating higher level of burden
Post-COVID-19 functional status (self-reported) | Week 10
  Post-COVID-19 Functional Status Scale - Patient Version (PCFS): self-report scale from 0 - 4 points with 0 = no functional limitations and 4 = severe functional limitations
Post-COVID-19 functional status (self-reported) | Week 16
  Post-COVID-19 Functional Status Scale - Patient Version (PCFS): self-report scale from 0 - 4 points with 0 = no functional limitations and 4 = severe functional limitations
Health-related quality of life | Week 10
  Short-form Health Survey (SF-12): self-report scale from 0 - 100 with higher score indicates a better health state
Health-related quality of life | Week 16
  Short-form Health Survey (SF-12): self-report scale from 0 - 100 with higher score indicates a better health state
Fatigue | Week 10
  Chalder fatigue-scale (CFS): self-report scale from 0 - 33 points with higher scores indicating higher level of physical and mental fatigue
Fatigue | Week 16
  Chalder fatigue-scale (CFS): self-report scale from 0 - 33 points with higher scores indicating higher level of physical and mental fatigue
Anxiety and depression | Week 10
  Hospital Anxiety and Depression Scale (HADS): self-report scale form 0 - 42 with higher scores indicating higher levels of anxiety and depression
Anxiety and depression | Week 16
  Hospital Anxiety and Depression Scale (HADS): self-report scale form 0 - 42 with higher scores indicating higher level of anxiety and depression
Insomnia | Week 16
  Insomnia Severity Index (ISI): self-report scale from 0 - 28 points with higher score indicating higher level of insomnia
Insomnia | Week 10
  Insomnia Severity Index (ISI): self-report scale from 0 - 28 points with higher score indicating higher level of insomnia
Cardiovascular performance | Week 10
  6-Minute-Walking-Test (6MWT): a longer traveled distance indicates a higher level of cardiovascular/pulmonary capacity
Cardiovascular performance | Week 16
  6-Minute-Walking-Test (6MWT): a longer traveled distance indicates a higher level of cardiovascular/pulmonary capacity
Pulmonary performance | Week 10
  Borg Breathlessness Scale (Borg-CR10-Scale): scale from 0-10 with higher scores indicating higher breathlessness/dyspnea - assesed subsequent to the 6-Minute-Walking-Test
Pulmonary performance | Week 16
  Borg Breathlessness Scale (Borg-CR10-Scale): scale from 0-10 with higher scores indicating higher breathlessness/dyspnea - assesed subsequent to the 6-Minute-Walking-Test
Post-COVID-19 functional status (physician-reported) | Week 10
  Post-COVID-19 Functional Status Scale - Physician Version (PCFS): physician-report scale from 0 - 4 points with 0 = no functional limitations and 4 = severe functional limitations
Post-COVID-19 functional status (physician-reported) | Week 16
  Post-COVID-19 Functional Status Scale - Physician Version (PCFS): physician-report scale from 0 - 4 points with 0 = no functional limitations and 4 = severe functional limitations
Adverse events | Weeks 0 - 10
  All adverse events in relation and unrelated to the intervention

OTHER OUTCOMES:
Treatment Expectation | Week 0
  Treatment Credibility Scale (TCS): expectation about the treatment effectiveness measured from 0 = no effectiveness to 10 = highest possible effectiveness
Self-efficacy | Week 10
  Arthritis Self-Efficacy Scale (ASES): the scale ranges from 1 to 10 with higher scores indicating more perceived efficacy
Self-efficacy | Week 16
  Arthritis Self-Efficacy Scale (ASES): the scale ranges from 1 to 10 with higher scores indicating more perceived efficacy
Stress | Week 10
  Perceived Stress Scale (PSS): 10-item scale, summed to create a psychological stress score of maximal 40 points with higher scores indicating greater psychological stress
Stress | Week 16
  Perceived Stress Scale (PSS): 10-item scale, summed to create a psychological stress score of maximal 40 points with higher scores indicating greater psychological stress
Flourishing | Week 10
  Flourishing-Scale (FS): the scale ranges from 8 (lowest possible value) to 56 (highest possible value) with higher values correspond to a person with many psychological resources and strengths
Flourishing | Week 16
  Flourishing-Scale (FS): the scale ranges from 8 (lowest possible value) to 56 (highest possible value) with higher values correspond to a person with many psychological resources and strengths
Loneliness | Week 10
  UCLA Loneliness Scale (UCLA-LS): the short form of the UCLA-LS constsis of 12 items, ranges from 0 to 36 points, with higher higher scores indicating greater loneliness
Loneliness | Week 16
  UCLA Loneliness Scale (UCLA-LS): the short form of the UCLA-LS constsis of 12 items, ranges from 0 to 36 points, with higher higher scores indicating greater loneliness

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof. MD, Study Chair — University of Duisburg-Essen; Heidemarie Haller, PhD, Principal Investigator — University of Duisburg-Essen; Christoph Kleinschnitz, Prof. MD, Study Director — University of Duisburg-Essen; Mark Stettner, Prof. MD, Study Director — University of Duisburg-Essen
Locations (1):
- Center for Integrative Medicine and Planetary Health, University Hospital Essen, University of Duisburg-Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No